CLINICAL TRIAL: NCT04578353
Title: Evaluation of the Safety & Performance of the AquaPass Medical Device, for Enhancing Fluid Transfer Through the Skin, by Increased Sweat Rate, on Healthy Volunteers and Chronic Edematous Patients
Brief Title: Effect of Enhanced Sweat Rate on the Safety and Edema Status of Chronic Edematous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AquaPass Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-003-01
Record Dates: First submitted 2020-09-25; First posted 2020-10-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-08

CONDITIONS: Chronic Heart Failure
Keywords: CHF; Edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AquaPass System (Experimental): Participants will undergo 3 procedures (each procedure up to 3 (±1) hours operation) using the AquaPass System, with 4-10 days between each procedure.
  Interventions: Device: The AquaPass System

INTERVENTIONS:
Device: The AquaPass System — The AquaPass device is a capsule that creates relatively homogenous temperature around the patients' lower body, while controlling and maintaining at a low percentage the relative humidity within the capsule thus enabling controlled environment that enhances sweat rate.

SUMMARY:
The purpose of this study is to demonstrate safety and performance of AquaPass System for enhancing fluid transfer through the skin, by increased sweat rate, in edematous patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, open label single arm study, conducted in two phases: up to 6 healthy subjects (Phase 1) and up to 16 chronic heart failure (CHF) patients (Phase 2).

After being informed about the study, requirements and potential risks, consenting patients will be enrolled and undergo 3 procedures (each procedure up to 3 (±1) hours operation), with 4-10 days between each procedure.

All patients will be followed up for 7 (±2) days from final procedure.

ELIGIBILITY:
Inclusion Criteria:

Phase 1: Healthy subjects:

1. Age ≥ 18
2. Subject has been informed on the nature of the study and has provided informed consent
3. Subject is capable of meeting study requirements

Phase 2: CHF Patients:

1. Age ≥ 18 and diagnosed with CHF
2. Subject has 2 or more score for pitting edema
3. Subject is taking diuretic medications at home
4. Subject has been informed on the nature of the study and has provided informed consent
5. Subject is capable of meeting study requirements

Exclusion Criteria:

Phase 1: Healthy subjects:

1. Subject is enrolled to another clinical investigation that might interfere with this study
2. Subject is pregnant or planning to become pregnant within the study period, or lactating mothers
3. Subject has no known sensitivity to Neoprene

Phase 2: CHF Patients:

1. Subject is enrolled to another clinical investigation that might interfere with this study
2. Subject is admitted to the hospital for acute decompensated or acute heart failure
3. Subject has any known lower body skin problems (open wounds, ulcers)
4. eGFR<15 ml/min/m2
5. Subject with severe peripheral arterial disease
6. Subject is pregnant or planning to become pregnant within the study period, or lactating mothers
7. Subject has known sensitivity to Neoprene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Safety Events | 30 days
  Device related SAE
System Activation | During procedure
  Ability to activate the AquaPass System and control skin temperature to levels between 33°C and 38°C
Treatment Toleration | During procedure
  Subjects can tolerate at least 2 hours of treatment

OTHER OUTCOMES:
Skin Changes | Before and and immediately after procedure
  Signs of burns grade 1 or more
CBC | Before and and immediately after procedure
  Change in Complete Blood Count
NT-proBNP (phase 2 only) | Before and and immediately after procedure
  Change in N-terminal prohormone of brain natriuretic peptide levels
Serum creatinine, BUN and Sodium | Before and and immediately after procedure
  Change in serum creatinine, blood urea nitrogen (BUN) and sodium levels
Urinary sodium concentration | Before and and immediately after procedure
  Change in urinary sodium concentration
Dyspnea | Before and and immediately after procedure
  Change in dyspnea score
Pitting edema | Before and and immediately after procedure
  Change in pitting edema score
JVD | Before and and immediately after procedure
  Change in jugular venous distention (JVD) score
Weight | During and and immediately after procedure
  Changes in weight

CONTACTS AND LOCATIONS:
Overall Officials: Doron Aronson, Professor, Principal Investigator — (Director, Inpatient Cardiology Unit (Rambam Health Care Campus)
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aronson D, Nitzan Y, Petcherski S, Bravo E, Habib M, Burkhoff D, Abraham WT. Enhancing Sweat Rate Using a Novel Device for the Treatment of Congestion in Heart Failure. Circ Heart Fail. 2023 Jan;16(1):e009787. doi: 10.1161/CIRCHEARTFAILURE.122.009787. Epub 2022 Nov 2. PMID 36321445